CLINICAL TRIAL: NCT04455373
Title: Long-term Outcome in Pediatric Surgical Bypass Grafting After Traumatic Injury and Tumor Resection
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stephanie Kampf, MD, Long-term outcome in pediatric surgical bypass grafting after traumatic injury and tumor resection, Medical University of Vienna
Other Study IDs: 1025/2018
Record Dates: First submitted 2020-06-23; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Child Health; Bypass Graft Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- orthopedic surgery group: Planned tumor resection
  Interventions: Procedure: pediatric vascular bypass grafting
- traumatic surgery group: Patients with traumatic vascular injury
  Interventions: Procedure: pediatric vascular bypass grafting

INTERVENTIONS:
Procedure: pediatric vascular bypass grafting — pediatric vascular bypass grafting

SUMMARY:
Introduction:

Vascular bypass surgery in children differs significantly from adults. It is a rarely performed procedure in the setting of trauma and tumor surgery to facilitate limb salvage. Beside the technical challenges to reconstruct the small and spastic vessels, bypass grafting should not impede growth of the extremity. The primary aim of this study was to assess long-term outcome after pediatric bypass grafting, in a single academic center, focusing on potential effects on limb development.

Methods:

In this retrospective cohort analyses we included all pediatric patients undergoing vascular bypass grafting at the Medical University of Vienna between 2002-2017. All patients ≤ 18 years suffered a traumatic injury or underwent a tumor resection of the lower or upper limb, respectively. The youngest female patient was 0.4 years, the youngest male patient was 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* age <18 years
* planned vascular bypass grafting

Exclusion Criteria:

* age >18 years
* no vascular intervention

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study represents a retrospective cohort analysis of pediatric patients who underwent vascular bypass grafting by an experienced team of vascular surgeons at the Medical University Vienna between 2002-2017.
  All data regarding demographics, operative techniques and outcome were collected from the in-hospital database registry in collaboration with the Department of Orthopedics and Trauma-Surgery. All patients ≤ 18 years who suffered a traumatic injury or vascular surgery due to a planned orthopedic extremity tumor resection were included in this study. 33 patients underwent vascular repair, a total of 15 patients fulfilling the criteria could be identified.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
bypass growth | 10 years
  bypass growth

SECONDARY OUTCOMES:
autologous vs. PTFE graft | patency rate in 1 year
  patients will either receive an autologous bypass graft or PTFE graft
revision surgery | <30 days
  revision surgery

IPD SHARING:
Plan to Share IPD: No